CLINICAL TRIAL: NCT00378053
Title: A Prospective Study of Radiation Exposure to Surgeons
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Other Study IDs: 060829
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2007-08

CONDITIONS: Radiation Exposure
Keywords: Radiation; Exposure; Hand; Orthopaedic; Surgeons

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to measure the amount of radiation over a specific period of time that Orthopaedic Surgeons are exposed to while using the mini c-arm fluoroscopy machine.

DETAILED DESCRIPTION:
The purpose of this study is to measure the amount of radiation over a specific period of time that Orthopaedic Surgeons are exposed to while using the mini c-arm fluoroscopy machine. The amount of radiation that the Surgeons will be exposed to will be recorded by a ring dosimeter located on the Surgeons' hand, and two badge dosimeters (one above the scrub collar, and one underneath a lead gown at waist level).

ELIGIBILITY:
This study will only enroll the Surgeons of the Vanderbilt Hand and Upper Extremity Center. There will be no inclusion/exclusion criteria for the type of surgery that will be monitored, nor the patients that are having surgery. If a mini c-arm fluoroscopy is used the amount of radiation received by the Surgeon's hand for that surgery will be monitored by a gas-sterilized radiation ring dosimeter. The amount of scatter radiation the Surgeon will be exposed to will be recorded by a badge dosimeter located on the Surgeon's scrub collar, and one badge dosimeter that will be located under the required lead gown worn by the Surgeon.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4
Dates: Start 2006-09; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Lee, M.D., Principal Investigator — VUMC
Locations (1):
- Vanderbilt University Medical Center- Vanderbilt Orthopaedic Institute, Nashville, Tennessee, United States